CLINICAL TRIAL: NCT05912244
Title: A Phase II Study of IO102/IO103 and Nivolumab-relatlimab Fixed Dose Combination in Untreated, Unresectable Stage III/IV Melanoma
Brief Title: A Study of IO102/IO103, Nivolumab, and Relatlimab in People With Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: IO Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-098
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: IO102/IO103; Nivolumab; Relatlimab; Unresectable; Stage III/IV; 23-098
MeSH Terms: conditions — Melanoma | interventions — Opdualag

STUDY DESIGN:
Intervention Model Description: Sequentially in a single-arm, nonrandomized two-stage trial design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IO102/IO103, Nivolumab, and Relatlimab (Experimental): All patients will be treated with nivolumab-relatlimab FDC on Day 1 of every 28-day cycle for up to two years. Patients will be treated with IO102/IO103 on Days 1 and 15 of the first two 28-day cycles, then on Day 1 of subsequent cycles for up to two total years of treatment.
  Interventions: Drug: IO102/IO103; Drug: Nivolumab-Relatlimab

INTERVENTIONS:
Drug: IO102/IO103 — IO102/IO103 will be administered subcutaneously on Days 1 and 15 of the first two 28-day cycles, and then on Day 1 only of subsequent cycles for two total years of treatment. Each vaccine contains 85ug.
Drug: Nivolumab-Relatlimab — Nivolumab-relatlimab will be administered as a single infusion 160mg relatlimab and nivolumab 480 mg for all participants. Both agents will be combined in a single fixed-dose combination (FDC) as an intravenous 30-minute infusion every four weeks.

SUMMARY:
The researchers are doing this study to find out whether the study vaccines, IO102/IO103, given in combination with the standard-of-care drug combination, nivolumab and relatlimab, is a safe and effective treatment for people with untreated, unresectable melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent
2. Patient must be able to provide informed consent.
3. Patient must have a histologically confirmed diagnosis of locally advanced unresectable stage III or metastatic stage IV melanoma not amenable to local therapy.
4. Patient must have not received any prior systemic therapy directed against unresectable stage III or IV melanoma. Prior neoadjuvant and adjuvant ICIs and BRAF/MEK inhibitors are permitted as long as the last dose was > 6 months prior to recurrence.
5. Patients must have at least one extraskeletal, extracranial measurable melanoma lesion as defined by RECIST v1.1. Note: A formal RECIST read by a study radiologist is not needed at the time of enrollment. Measurable disease can be assessed by the treating investigator.
6. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
7. Adequate laboratory function at screening, defined as:

   1. Hemoglobin ≥ 9.0 g/dL
   2. WBC ≥ 2000/uL
   3. Platelet count ≥ 100 × 10^9 /L
   4. Serum direct bilirubin ≤ 1.5 × upper limit of normal (ULN); AST and ALT ≤ 2.5 × ULN. (Total bilirubin < 3 mg/dL for subjects with Gilbert's disease)
   5. Calculated creatinine clearance (CrCl) ≥15 mL/min based on the Cockcroft-Gault equation
8. Patients of childbearing potential* who are sexually activ partner must use two methods of effective contraception from screening, and must agree to continue using such precautions for 23 weeks after the final dose of investigational product: cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

   *Patients of childbearing potential are defined as those who are assigned female at birth and not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
9. Male patients who are sexually active with partners of childbearing potential must use highly effective methods of contraception throughout the study and for at least four months following the last dose of study treatment. Male patients must agree not to donate sperm during the study treatment period.

Exclusion Criteria:

1. Uveal melanoma
2. Untreated central nervous system (CNS) metastases or any leptomeningeal involvement. Asymptomatic brain metastases that have been treated with external radiotherapy are permitted.
3. Any immunotherapy treatment for unresectable stage III/IV melanoma or any other prior unresectable malignancy. Prior neoadjuvant and adjuvant ICIs and BRAF/MEK inhibitors are permitted as long as the last dose was > 6 months prior to recurrence.
4. Systemic steroid therapy higher than physiologic dose steroid replacement (>10 mg/day of prednisone or equivalent), given within 14 days of starting treatment, or other immunosuppressive medications within 14 days of the start of treatment. Inhaled or topical steroids are permitted in the absence of active autoimmune disease. 5. Treatment with any live/attenuated vaccine within 30 days of first study treatment. Inactivated and mRNA vaccines are permitted.

6. History of motor neuropathy considered to be of autoimmune origin to be of autoimmune origin (e.g., Guillain-Barre syndrome, myasthenia gravis) 7. Other active, concurrent malignancy that requires ongoing systemic treatment or interferes with radiographic assessment of melanoma response as determined by the investigator 8. History of severe allergic reactions to any unknown allergens or any components of the study drugs.

9. Uncontrolled (i.e., unstable) concomitant medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety or compliance with the study procedures. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. 10. Active hepatitis B virus (HBV) with a viral load >100 IU/mL 11. Active hepatitis C virus (HCV) with a viral load >100 IU/mL 12. Patients who are breastfeeding or who are pregnant as evidenced by a positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) performed within 14 days of the first dose of study drug.

13. Prisoners or participants who are involuntarily incarcerated. (Note: Under certain specific circumstances where local regulations permit, a person who has been imprisoned may be permitted to continue as a participant.) 14. Participants who are compulsorily detained for treatment of either a psychiatric or physical illness (e.g., transmissible infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 3 years
  will be reported as the proportion of patients who experience a complete (CR) or partial response (PR) to treatment by RECIST v1.1

SECONDARY OUTCOMES:
Incidence of adverse events | up to 100 days after the last dose
  graded and recorded according to CTCAE v5.0
Progression-free survival (PFS) | 3 years
  by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: James Smithy, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Hartford Healthcare Alliance (Data Collection Only), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Background] Kjeldsen JW, Lorentzen CL, Martinenaite E, Ellebaek E, Donia M, Holmstroem RB, Klausen TW, Madsen CO, Ahmed SM, Weis-Banke SE, Holmstrom MO, Hendel HW, Ehrnrooth E, Zocca MB, Pedersen AW, Andersen MH, Svane IM. A phase 1/2 trial of an immune-modulatory vaccine against IDO/PD-L1 in combination with nivolumab in metastatic melanoma. Nat Med. 2021 Dec;27(12):2212-2223. doi: 10.1038/s41591-021-01544-x. Epub 2021 Dec 9. PMID 34887574
- [Background] Lorentzen CL, Kjeldsen JW, Ehrnrooth E, Andersen MH, Marie Svane I. Long-term follow-up of anti-PD-1 naive patients with metastatic melanoma treated with IDO/PD-L1 targeting peptide vaccine and nivolumab. J Immunother Cancer. 2023 May;11(5):e006755. doi: 10.1136/jitc-2023-006755. PMID 37217243
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm